CLINICAL TRIAL: NCT00010530
Title: Basic Mechanisms of Meditation and Cardiovascular Disease in Older Blacks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: P50AT000082-01P1 (NIH); P50AT000082-01 (NIH); P50AT000082-02 (NIH); NCT00009087 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Cardiovascular Diseases
Keywords: CVD
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Meditation

SUMMARY:
The purpose of this study is to evaluate the effects of meditation on older African Americans with documented cardiovascular disease (CVD).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death and disability in older African Americans, and accounts for 40% of the disproportionate risk for mortality observed in African Americans compared to white Americans. The majority of CVD patients experience acute cardiac events, many sudden and unexpected, despite conventional treatment of their disease and associated traditional risk factors. The pathophysiologic basis of these cardiac events is not fully established, but substantial evidence indicates that psychosocial stress and the sympathetic nervous system have adverse effects on both vasomotor function and long-term autonomic balance. Recent advances in the understanding of the pathophysiology of acute cardiac events-specifically, the roles that arterial vasomotor dysfunction and sympathetic nervous system imbalance play in the pathophysiology of such acute events-provide a platform for a new mechanistic investigation of the interplay of psychosocial and environmental stress and CVD. Preliminary evidence demonstrating elevated peripheral vasoconstriction due to stress-mediated sympathetic nervous system response in African Americans further suggests that these mechanisms are particularly relevant in this group.

ELIGIBILITY:
Inclusion Criteria:

* African-American (self-identified)
* Local residence
* Able to participate
* Coronary artery disease by MI, CABG, PTCA (>3 months prior), or angiography
* Consent and referring MD approval

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1999-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Schneider, MD, Principal Investigator — Center for Health and Aging Studies
Locations (2):
- United States (2):
  - Charles R. Drew University of Medicine and Science, Los Angeles, California
  - Maharishi University of Management Center for Health and Aging Studies, Fairfield, Iowa